CLINICAL TRIAL: NCT03250442
Title: A Randomized Controlled Trial Evaluating the Outcomes for Incisional Application of Negative Pressure for Nontraumatic Lower Extremity Amputations: A Pilot Study
Brief Title: Evaluating the Outcomes for Incisional Application of Negative Pressure for Nontraumatic Amputations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0599
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Surgical Wound; Wound Heal; Amputation
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A: Standard Dry Dressing (Other): The standard dry dressing is comprised of nonadherent dressing, dry gauze, cotton undercast padding, compression, and immobilization.
  Interventions: Other: Standard Dry Dressing
- Group B: Foam, Drape, and PrevenaTM (Active Comparator): This arm is comprised of foam, drape, the PrevenaTM Device, compression, and immobilization.
  Interventions: Device: PrevenaTM Device

INTERVENTIONS:
Device: PrevenaTM Device — The PrevenaTM Incision Management System covers and protects the incision from external contamination, while negative pressure removes fluid and infectious material from the surgical incision.
  Arms: Group B: Foam, Drape, and PrevenaTM
Other: Standard Dry Dressing — These are customary dry dressings.
  Arms: Group A: Standard Dry Dressing

SUMMARY:
The purpose of this study is to evaluate how well subjects heal after surgery who receive standard dressings or incisional negative pressure wound therapy for non-traumatic amputation sites.

DETAILED DESCRIPTION:
Incisional negative pressure wound therapy is an approved device used for wound healing of closed surgical incisions. This research is being done because incisional negative pressure wound therapy is a new application of negative pressure wound therapy that is applied over a closed incision area instead of an open wound. Negative pressure wound therapy is commonly used to help heal open wounds. It involves the use of a piece of foam, an adhesive drape, and a battery-powered device that places negative pressure on the wound. Currently, there are no trials utilizing incisional negative pressure wound therapy of closed wounds after below knee amputations (BKA), transmetatarsal amputations (TMA), Knee Disarticulations (KD), and Above Knee Amputations (AKA). This is a pilot study that compares incisional negative pressure wound therapy and standard dressings in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years or older to participate.
2. Requires closure of a nontrauamtic Transmetatarsal Amputation (TMA), Below Knee Amputation (BKA), Knee Disarticulation (KD), or Above Knee Amputation (AKA).
3. Has at least one artery that feeds the closure site.
4. Able to comply with clinical trial procedures and schedule.

Exclusion Criteria:

1. Patients not receiving an amputation.
2. The investigator/provider determines that the patient has an indication against incisional negative pressure wound therapy that would prevent them from participating.
3. Surgical incision that is not completely closed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of postoperative incision complications between the 2 arms | 95 days
  The proportion of issues that arise between the two groups after closure surgery.

SECONDARY OUTCOMES:
Length of hospital stay | 5 days
  The amount of time the patients must stay after closure surgery.
Number of surgically related wound readmissions | 95 days
  The number of times patients are readmitted to the hospital for their surgical wound post-discharge.
Medical Outcomes Study 12 Short Form Health Survey (SF-12) | 95 days
  Change in quality of life from the start of the study to the end.
Percentage of closed incisions remained closed at 1, 2 and 3 months post-hospital discharge | At 1, 2, and 3 months post-hospital discharge
  The percentage of closed surgical wounds that remain closed after 1, 2 and 3 months after their closure surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Attinger, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No